CLINICAL TRIAL: NCT02639546
Title: A Phase I/II, Multicenter, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of Cobimetinib In Pediatric and Young Adult Patients With Previously Treated Solid Tumors
Brief Title: Safety and Pharmacokinetics of Cobimetinib in Pediatric and Young Adult Participants With Previously Treated Solid Tumors
Acronym: iMATRIXcobi
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO29665; 2014-004685-25 (EudraCT Number)
Record Dates: First submitted 2015-12-03; First posted 2015-12-24 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Solid Tumors
MeSH Terms: interventions — cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase I (Tablet) Cobimetinib (0.6 mg/kg) (Experimental): Dose-Escalation: Participants received 0.6 milligrams per kilogram (mg/kg) cobimetinib orally once daily on Days 1 to 21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib
- Phase I (Tablet) Cobimetinib (0.8 mg/kg) (Experimental): Dose-Escalation: Participants received 0.8 milligrams per kilogram (mg/kg) cobimetinib orally once daily on Days 1 to 21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib
- Phase I (Tablet) Cobimetinib (1 mg/kg) (Experimental): Dose-Escalation: Participants received 1 milligram per kilogram (mg/kg) cobimetinib orally once daily on Days 1 to 21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib
- Phase I (Suspension) Cobimetinib (0.6 mg/kg) (Experimental): Dose-Escalation: Participants received 0.6 milligrams per kilogram (mg/kg) cobimetinib orally once daily on Days 1 to 21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib
- Phase I (Suspension) Cobimetinib (0.8 mg/kg) (Experimental): Dose-Escalation: Participants received 0.8 milligrams per kilogram (mg/kg) cobimetinib orally once daily on Days 1 to 21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib
- Phase I (Suspension) Cobimetinib (1 mg/kg) (Experimental): Dose-Escalation: Participants received 1 milligram per kilogram (mg/kg) cobimetinib orally once daily on Days 1 to 21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib
- Phase I (Suspension) Cobimetinib (1.33 mg/kg) (Experimental): Dose-Escalation: Participants received 1.33 milligrams per kilogram (mg/kg) cobimetinib orally once daily on Days 1 to 21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib
- Phase II (Suspension) Cobimetinib (1 mg/kg) (Experimental): Dose-Expansion: Participants received 1 milligram per kilogram (mg/kg) cobimetinib orally once daily on Days 1 to 21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib tablet or suspension will be administered as per the schedule described in arm description.
  Other Names: RO5514041, GDC-0973, XL-518

SUMMARY:
This open-label, dose-escalation study is designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of cobimetinib in pediatric and young adult participants with solid tumors with known or potential kinase pathway activation for which standard therapy has proven to be ineffective or intolerable or for which no curative standard-of-care treatment options exist. The study will be conducted in two stages: a dose-escalation stage and an expansion stage at the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* For dose-escalation stage (tablets): age at study entry >= 6 years to < 18 years
* For dose-escalation stage (suspension): age at study entry >= 6 months to < 18 years. Participants <1 year of age will not be enrolled until >= 6 participants >= 1 year to < 18 years of age have received at least one cycle of therapy with suspension and until safety and pharmacokinetic assessment of these participants have been conducted.
* For expansion stage: age at study entry to be >= 6 months (>=6 years if suspension is not available) to < 30 years. Participants >= 6 months to < 1 year of age may not be enrolled until >= 6 participants >= 1 year to < 18 years of age have received at least one cycle of therapy with suspension in the dose-escalation phase and until safety and pharmacokinetic assessment of these participants have been conducted.
* Tumor for which prior treatment has proven to be ineffective or intolerable or for which no standard therapy exists
* Tumor with known or expected RAS/RAF/MEK/ERK pathway involvement. Diagnosis must be one of the following tumor types:

Central nervous system gliomas, including high- and low-grade gliomas, and diffuse intrinsic pontine glioma (DIPG) Embryonal rhabdomyosarcoma and other non-rhabdomyosarcoma soft tissue sarcomas Neuroblastoma Melanoma Malignant peripheral nerve sheath tumor Rhabdoid tumors, including atypical teratoid/rhabdoid tumor (ATRT) NF1-associated tumor (including plexiform neurofibroma), schwannoma, or RASopathy-associated tumor that in the judgment of the investigator is life threatening, results in severe symptoms (including severe pain), or is in close proximity to vital structures

* Measurable disease as defined by mINRC, RANO criteria for HGG, RANO criteria for LGG, RECIST v1.1, or evaluable by nuclear medicine techniques, immunocytochemistry, tumor markers, or other reliable measures
* Availability of tumor tissue at study enrollment
* Lansky performance status or Karnofsky performance status of >= 50 percent
* Life expectancy >= 3 months
* Adequate hematologic, cardiac, and end-organ function
* Body weight must be >= 20 kilograms (kg) if suspension is not available

Exclusion Criteria:

* Pregnant or lactating women
* Close proximity in time to treatment with high-dose chemotherapy, stem-cell rescue, differentiation therapy, immunotherapy, thoracic or mediastinal radiotherapy, hormonal therapy, biologic therapy, herbal cancer therapy, hematopoietic growth factor, investigational therapy, or St. John's wort according to protocol-defined criteria prior to initiation of study drug
* Inability to swallow oral medications
* Impaired gastrointestinal absorption
* History or evidence of retinal pathology according to protocol-defined criteria, including serous retinopathy
* History of Grade >= 2 central nervous system (CNS) hemorrhage
* History of CNS hemorrhage within 28 days of study entry. This criterion may be waived at the investigator's request if the CNS hemorrhage was asymptomatic, with approval of the Medical Monitor
* Known active infection (excluding fungal infection of the nail beds) within 28 days prior to initiation of study drug that has not completely resolved
* Major surgical procedure or significant traumatic injury within 4 weeks prior to initiation of study drug, or anticipation of need for major surgical procedure during the course of the study
* Prior allogenic bone marrow transplantation or prior solid organ transplantation

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (5):
  - Arkansas Children'S Hospital, Little Rock, Arkansas
  - Arnold Palmer Hosp-Children, Orlando, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- France (3):
  - Hôpital de la Timone, Oncologie Pédiatrique, Marseille
  - Institut Curie, Oncologie Pédiatrique, Paris
  - Institut Gustave Roussy; Service Pediatrique, Villejuif
- Universitaetsklinikum Muenster, Münster, Germany
- Schneider Children's Medical Center, Petah Tikva, Israel
- Fondazione IRCCS Istituto Nazionale dei Tumori; Struttura Complessa di Pediatria Oncologica, Milan, Lombardy, Italy
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- United Kingdom (3):
  - Alderhey Childrens Trust, Liverpool
  - Great Ormond Street Hospital; Dept. Of Pediatric Oncology, London
  - The Royal Victoria Infirmary; Paediatric and Adolescent Oncology Unit, Newcastle upon Tyne

REFERENCES:
- [Derived] Trippett T, Toledano H, Campbell Hewson Q, Verschuur A, Langevin AM, Aerts I, Howell L, Gallego S, Rossig C, Smith A, Patel D, Pereira LR, Cheeti S, Musib L, Hutchinson KE, Devlin C, Bernardi R, Geoerger B. Cobimetinib in Pediatric and Young Adult Patients with Relapsed or Refractory Solid Tumors (iMATRIX-cobi): A Multicenter, Phase I/II Study. Target Oncol. 2022 May;17(3):283-293. doi: 10.1007/s11523-022-00888-9. Epub 2022 Jun 17. PMID 35715627

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 centers in 7 countries.
Pre-assignment Details: A total of 63 participants were screened, of which a total of 56 participants were enrolled. Tumor type was not a determinant of cohort assignment for the phase I portion of the study. The phase II portion of the study was restricted to participants with Low-Grade Glioma.
Period: Overall Study
Arm/Group | Phase I (Tablet) Cobimetinib (0.6 mg/kg) | Phase I (Tablet) Cobimetinib (0.8 mg/kg) | Phase I (Tablet) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (0.6 mg/kg) | Phase I (Suspension) Cobimetinib (0.8 mg/kg) | Phase I (Suspension) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (1.33 mg/kg) | Phase II (Suspension) Cobimetinib (1 mg/kg)
Started | 6 | 6 | 6 | 6 | 7 | 8 | 5 | 12
Tumor Type - Neuroblastoma | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumor Type - High-Grade Glioma | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tumor Type - Low-Grade Glioma | 1 | 2 | 4 | 5 | 3 | 2 | 3 | 12
Tumor Type - Dnet In Noonan's Syndrome Tumor With RAS/RAF/MEK/ERK Pathway Activation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumor Type - Malignant Peripheral Nerve Sheath Tumor | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tumor Type - Metastatic Mediastinal Yolksac Tumor With RAS/RAF/MEK/ERK Pathway Activation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumor Type - Non-Rhabdomyosarcoma Soft Tissue Sarcoma | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumor Type - Plexiform Neurofibroma | 1 | 2 | 1 | 1 | 2 | 4 | 1 | 0
Tumor Type - Rhabdoid Tumor/ATRT | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 6 | 7 | 8 | 5 | 12
Not completed — Death | 2 | 2 | 1 | 2 | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Not completed — PI, physician decision; no response to trt. | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Study Terminated By Sponsor | 0 | 2 | 3 | 4 | 4 | 3 | 3 | 9
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 0 | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I (Tablet) Cobimetinib (0.6 mg/kg) | Phase I (Tablet) Cobimetinib (0.8 mg/kg) | Phase I (Tablet) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (0.6 mg/kg) | Phase I (Suspension) Cobimetinib (0.8 mg/kg) | Phase I (Suspension) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (1.33 mg/kg) | Phase II (Suspension) Cobimetinib (1 mg/kg) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 5 | 12 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.8 (3.5) | 9.5 (3.3) | 9.5 (3.4) | 8.5 (1.4) | 9.7 (5.3) | 8.9 (3.1) | 10.2 (3.3) | 8.7 (7.5) | 9.5 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 2 | 0 | 2 | 5 | 7 | 23
  Male | 5 | 4 | 2 | 4 | 7 | 6 | 0 | 5 | 33
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 4 | 11
  Not Hispanic or Latino | 5 | 3 | 4 | 1 | 2 | 4 | 3 | 7 | 29
  Not Stated | 0 | 0 | 2 | 3 | 1 | 2 | 0 | 0 | 8
  Unknown | 0 | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Unknown | 1 | 1 | 2 | 5 | 4 | 3 | 1 | 1 | 18
  White | 5 | 4 | 3 | 0 | 2 | 5 | 4 | 11 | 34
Tumor Type [Count of Participants; unit: Participants]
  Neuroblastoma | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  High-Grade Glioma | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 5
  Low-Grade Glioma | 1 | 2 | 4 | 5 | 3 | 2 | 3 | 12 | 32
  Dnet In Noonan's Syndrome Tumor With RAS/RAF/MEK/ERK Pathway Activation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Malignant Peripheral Nerve Sheath Tumor | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Metastatic Mediastinal Yolksac Tumor With RAS/RAF/MEK/ERK Pathway Activation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Non-Rhabdomyosarcoma Soft Tissue Sarcoma | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Plexiform Neurofibroma | 1 | 2 | 1 | 1 | 2 | 4 | 1 | 0 | 12
  Rhabdoid Tumor/ATRT | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose-Limiting Toxicities (DLTs)
Description: Dose-Limiting Toxicities (DLTs) were defined as cobimetinib-related adverse events occurring within the first 28 days of each administration of cobimetinib.
Time Frame: Baseline up until 30 days after the last dose of study drug (up to 5 years, 2 months)
Population: The safety evaluable population was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase I (Tablet) Cobimetinib (0.6 mg/kg) | Phase I (Tablet) Cobimetinib (0.8 mg/kg) | Phase I (Tablet) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (0.6 mg/kg) | Phase I (Suspension) Cobimetinib (0.8 mg/kg) | Phase I (Suspension) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (1.33 mg/kg) | Phase II (Suspension) Cobimetinib (1 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 5 | 12
Percentage of Participants | 0 | 0 | 33.3 | 16.7 | 0 | 0 | 60.0 | 0

2. Primary Outcome: Percentage of Participants With Adverse Events (AEs), Including Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs.
Time Frame: Baseline up until 30 days after the last dose of study drug (up to 5 years, 2 months)
Population: The safety evaluable population was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase I (Tablet) Cobimetinib (0.6 mg/kg) | Phase I (Tablet) Cobimetinib (0.8 mg/kg) | Phase I (Tablet) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (0.6 mg/kg) | Phase I (Suspension) Cobimetinib (0.8 mg/kg) | Phase I (Suspension) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (1.33 mg/kg) | Phase II (Suspension) Cobimetinib (1 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 5 | 12
Percentage of Participants
  AEs | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  SAEs | 33.3 | 33.3 | 33.3 | 33.3 | 14.3 | 25.0 | 40.0 | 41.7
  AESIs | 33.3 | 33.3 | 33.3 | 50.0 | 42.9 | 25.0 | 100.0 | 58.3

3. Primary Outcome: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of Cobimetinib
Description: A prior dose level was defined as an MTD/MAD if at a certain dose level, there were greater than or equal to (>=) 2 out of 6 participants who had Dose Limiting Toxicities (DLTs).
Time Frame: Cycle 1 Day 1 up to Cycle 1 Day 28 (cycle length=28 days)
Population: The safety evaluable population was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: mg/kg
Groups:
- Cobimetinib (Tablet) Population: Participants received Cobimetinib (Tablet) formulation
- Cobimetinib (Suspension) Population: Participants received Cobimetinib (Suspension) formulation
Arm/Group | Cobimetinib (Tablet) Population | Cobimetinib (Suspension) Population
Number analyzed (Participants) | 18 | 38
mg/kg | 0.8 | 1

4. Primary Outcome: Percentage of Participants With Objective Response (Complete Response (CR) or Partial Response (PR)) as Determined by the Investigator Using Modified International Neuroblastoma Response Criteria (mINRC) for Participants With Neuroblastoma (Phase I)
Description: Tumor assessment was performed using mINRC for Participants with Neuroblastoma.
Time Frame: Baseline up to disease progression or death due to any cause, whichever occurs first (up to 5 years, 2 months)
Population: The safety evaluable population was defined as all participants who received at least one dose of study drug. Participants enrolled into phase I (Dose-Escalation) cohorts independent of their tumor type. As the same criteria were not used to assess response in all tumor types, the efficacy analyses were broken down by tumor type.
Measure: Number; unit: Percentage of Participants
Groups:
- Neuroblastoma: Participants with Neuroblastoma.
Arm/Group | Neuroblastoma
Number analyzed (Participants) | 1
Percentage of Participants | 0

5. Primary Outcome: Percentage of Participants With Objective Response (CR or PR) as Determined by the Investigator Using RANO Criteria for Participants With High-Grade Glioma (HGG) (Phase I) and RECIST v1.1 for Participants With Low-Grade Glioma (LGG) (Phase I and II)
Description: Tumor assessment was performed using Response Assessment in Neuro-Oncology (RANO) criteria for participants with HGG and Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) for participants with LGG. While the data for LGG in the phase II cohort is presented separately in other parts of the record, it was also considered useful to combine the data for LGG from phase I and phase II, which was done here.
Time Frame: Baseline up to disease progression or death due to any cause, whichever occurs first (up to 5 years, 2 months)
Population: The safety evaluable population was defined as all participants who received at least one dose of study drug. Participants enrolled into phase I (Dose-Escalation) cohorts independent of their tumor type. For phase II, only one tumor type cohort was opened (LGG). As the same criteria were not used to assess response in all tumor types, the efficacy analyses were broken down by tumor type.
Measure: Number; unit: Percentage of Participants
Groups:
- High Grade Glioma: Participants with High Grade Glioma.
- Low Grade Glioma: Participants with Low Grade Glioma.
Arm/Group | High Grade Glioma | Low Grade Glioma
Number analyzed (Participants) | 5 | 32
Percentage of Participants | 0 | 9.4

6. Primary Outcome: Percentage of Participants With Objective Response (CR or PR) as Determined by the Investigator Using RECIST v1.1 Criteria for Participants With All Other Tumours (Phase I)
Description: Tumor assessment was performed using RECIST v1.1 for Participants with All Other Tumours.
Time Frame: Baseline up to disease progression or death due to any cause, whichever occurs first (up to 5 years, 2 months)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Groups:
- Dnet In Noonan's Syndrome Tumor With RAS/RAF/MEK/ERK Pathway Activation: Participants with Dnet In Noonan's Syndrome Tumor With RAS/RAF/MEK/ERK Pathway Activation.
- Malignant Peripheral Nerve Sheath Tumor: Participants with Malignant Peripheral Nerve Sheath Tumor.
- Metastatic Mediastinal Yolksac Tumor With RAS/RAF/MEK/ERK Pathway Activation: Participants with Metastatic Mediastinal Yolksac Tumor With RAS/RAF/MEK/ERK Pathway Activation.
- Non-Rhabdomyosarcoma Soft Tissue Sarcoma: Participants with Non-Rhabdomyosarcoma Soft Tissue Sarcoma.
- Plexiform Neurofibroma: Participants with Plexiform Neurofibroma.
- Rhabdoid Tumor/ATRT: Participants with Rhabdoid Tumor/ATRT.
Arm/Group | Dnet In Noonan's Syndrome Tumor With RAS/RAF/MEK/ERK Pathway Activation | Malignant Peripheral Nerve Sheath Tumor | Metastatic Mediastinal Yolksac Tumor With RAS/RAF/MEK/ERK Pathway Activation | Non-Rhabdomyosarcoma Soft Tissue Sarcoma | Plexiform Neurofibroma | Rhabdoid Tumor/ATRT
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 12 | 1
Percentage of Participants | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Percentage of Participants With Objective Response (CR or PR) as Determined by the Investigator Using RANO Criteria for Participants With LGG (Phase II)
Description: Tumor assessment will be performed using RANO criteria for LGG.
Time Frame: Baseline up to disease progression or death due to any cause, whichever occurs first (up to 5 years, 2 months)
Population: The safety evaluable population was defined as all participants who received at least one dose of study drug. For phase II, only one tumor type cohort was opened (LGG).
Measure: Number; unit: Percentage of Participants
Arm/Group | Low Grade Glioma
Number analyzed (Participants) | 12
Percentage of Participants | 8.3

8. Primary Outcome: Progression-Free Survival (PFS) as Determined by the Investigator Using mINRC for Participants With Neuroblastoma (Phase I)
Description: Tumor assessment was performed using mINRC for Participants with Neuroblastoma.
Time Frame: From the time of cobimetinib study drug initiation to the first documented disease progression, or death due to any cause, whichever occurs first (up to 5 years, 2 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Neuroblastoma
Number analyzed (Participants) | 1
Months | 1.3 [NA to NA] — The confidence interval could not be calculated from the data of one participant.

9. Primary Outcome: PFS as Determined by the Investigator Using RANO Criteria for Participants With HGG (Phase I) and RECIST v1.1 for Partcipants With LGG (Phase I and II)
Description: Tumor assessment was performed using RANO for participants with HGG and RECIST v1.1 for participants with LGG. While the data for LGG in the phase II cohort is presented separately in other parts of the record, it was also considered useful to combine the data for LGG from phase I and phase II, which was done here.
Time Frame: as for outcome 8
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | High Grade Glioma | Low Grade Glioma
Number analyzed (Participants) | 5 | 32
Months | 1.0 [0.6 to NA] — The upper limit could not be calculated from the data due to insufficient number of participants with events. | 22.0 [9.3 to NA] — The upper limit could not be calculated from the data due to insufficient number of participants with events.

10. Primary Outcome: PFS as Determined by the Investigator Using RECIST v1.1 Criteria for Participants With All Other Tumours (Phase I)
Description: Tumor assessment was performed using RECIST v1.1 for Participants with All Other Tumours.
Time Frame: as for outcome 8
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dnet In Noonan's Syndrome Tumor With RAS/RAF/MEK/ERK Pathway Activation | Malignant Peripheral Nerve Sheath Tumor | Metastatic Mediastinal Yolksac Tumor With RAS/RAF/MEK/ERK Pathway Activation | Non-Rhabdomyosarcoma Soft Tissue Sarcoma | Plexiform Neurofibroma | Rhabdoid Tumor/ATRT
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 12 | 1
Months | NA [NA to NA] — PFS could not be calculated from the data of 1 participant | 4.1 [0.7 to NA] — The upper limit could not be calculated from the data due to insufficient number of participants with events. | 1.1 [NA to NA] — The upper and lower limits could not be calculated from the data of 1 participant. | 3.4 [NA to NA] — The upper and lower limits could not be calculated from the data of 1 participant. | NA [18.4 to NA] — The upper limit could not be calculated from the data due to insufficient number of participants with events. | 0.5 [NA to NA] — The upper and lower limits could not be calculated from the data of 1 participant.

11. Primary Outcome: PFS as Determined by the Investigator Using RANO Criteria for Participants With LGG (Phase II)
Description: Tumor assessment was performed using RANO criteria for Participants with LGG.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Low Grade Glioma
Number analyzed (Participants) | 12
Months | 18.4 [3.6 to NA] — The upper limit could not be calculated from the data due to insufficient number of participants with events.

12. Secondary Outcome: Recommended Phase II Dose (RP2D) of Cobimetinib
Description: A prior dose level was defined as an RP2D if at a certain dose level, there were greater than or equal to (≥) 2 out of 6 participants who had Dose Limiting Toxicities (DLTs).
Time Frame: Cycle 1 Day 1 up to Cycle 1 Day 28 (cycle length=28 days)
Population: The safety evaluable population was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: mg/kg
Arm/Group | Cobimetinib (Suspension) Population
Number analyzed (Participants) | 38
mg/kg | 1

13. Secondary Outcome: Duration of Response (DOR) as Determined by the Investigator Using RECIST v1.1 for Participants With LGG (Phase I and II)
Description: Tumor assessment was performed using RECIST v1.1 criteria for participants with LGG. While the data for LGG in the phase II cohort is presented separately in other parts of the record, it was also considered useful to combine the data for LGG from phase I and phase II, which was done here.
Time Frame: From first occurrence of objective response to disease progression or death due to any cause, whichever occurs first (up to 5 years, 2 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Low Grade Glioma
Number analyzed (Participants) | 3
Months | NA [NA to NA] — No participants experienced an event and DOR was not reached.

14. Secondary Outcome: DOR as Determined by the Investigator RANO Criteria for Participants With LGG (Phase II)
Description: Tumor assessment was performed using RANO criteria for Participants with LGG.
Time Frame: as for outcome 13
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Low Grade Glioma
Number analyzed (Participants) | 1
Months | NA [NA to NA] — No participants experienced an event and DOR was not reached.

15. Secondary Outcome: Overall Survival (OS) for Participants With Neuroblastoma (Phase I)
Description: OS was defined as the time from initiation of study drug to death from any cause.
Time Frame: Baseline until death due to any cause (up to 5 years, 2 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Neuroblastoma
Number analyzed (Participants) | 1
Months | 4.6 [NA to NA] — The confidence interval could not be calculated from the data of one participant.

16. Secondary Outcome: OS for Participants With High-Grade Glioma (HGG) (Phase I) and Low-Grade Glioma (LGG) (Phase I and II)
Description: OS was defined as the time from initiation of study drug to death from any cause. While the data for LGG in the phase II cohort is presented separately in other parts of the record, it was also considered useful to combine the data for LGG from phase I and phase II, which was done here.
Time Frame: Baseline until death due to any cause (up to 5 years, 2 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | High Grade Glioma | Low Grade Glioma
Number analyzed (Participants) | 5 | 32
Months | 1.4 [0.6 to NA] — The upper limit cannot be calculated due to insufficient number of events. | NA [NA to NA] — No participants experienced an event and DOR was not reached.

17. Secondary Outcome: OS for Participants With All Other Tumours (Phase I)
Description: OS was defined as the time from initiation of study drug to death from any cause.
Time Frame: Baseline until death due to any cause (up to 5 years, 2 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dnet In Noonan's Syndrome Tumor With RAS/RAF/MEK/ERK Pathway Activation | Malignant Peripheral Nerve Sheath Tumor | Metastatic Mediastinal Yolksac Tumor With RAS/RAF/MEK/ERK Pathway Activation | Non-Rhabdomyosarcoma Soft Tissue Sarcoma | Plexiform Neurofibroma | Rhabdoid Tumor/ATRT
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 12 | 1
Months | NA [NA to NA] — The median and 95% confidence interval could not be calculated from the data of one participant. | 5.5 [0.8 to NA] — The upper limit could not be calculated from the data due to insufficient number of participants with events. | 1.1 [NA to NA] — The 95% confidence interval could not be calculated from the data of one participant. | 6.3 [NA to NA] — The 95% confidence interval could not be calculated from the data of one participant. | NA [NA to NA] — The median and 95% confidence interval could not be calculated from the data due to insufficient number of participants with events. | 5.1 [NA to NA] — The 95% confidence interval could not be calculated from the data of one participant.

18. Secondary Outcome: Maximum Plasma Concentration Observed (Cmax) of Cobimetinib
Description: Plasma samples for determination of Cobimetinib concentration were collected prior to dosing and at 2, 4, 6 and 24 hours after dosing on Days 1 and 21 of Cycle 1. The sampling will allow determination of Cmax.
Time Frame: Pre-dose, 2, 4, 6, and 24 hours post-dose on Cycle 1 Days 1 and 21 (predose=within 4 hours prior to dose; cycle length=28 days)
Population: The PK population was defined as all participants who received at least 1 dose of Cobimetinib and had evaluable PK data. Only participants for whom data were collected are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase I (Tablet) Cobimetinib (0.6 mg/kg) | Phase I (Tablet) Cobimetinib (0.8 mg/kg) | Phase I (Tablet) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (0.6 mg/kg) | Phase I (Suspension) Cobimetinib (0.8 mg/kg) | Phase I (Suspension) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (1.33 mg/kg) | Phase II (Suspension) Cobimetinib (1 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 5 | 12
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 5 | 6 | 6 | 7 | 8 | 4 | 9
  Cycle 1 Day 1 | 62.0 (82.3) | 88.3 (102) | 144 (58.6) | 51.5 (73.4) | 67.4 (165) | 136 (80.3) | 111 (37.0) | 44.0 (69.8)
  Cycle 1 Day 21: number analyzed (Participants) | 5 | 5 | 5 | 6 | 6 | 8 | 2 | 9
  Cycle 1 Day 21 | 51.1 (74.0) | 181 (134) | 193 (35.0) | 105 (84.5) | 156 (91.2) | 179 (113) | 172 (60.3) | 116 (42)

19. Secondary Outcome: Time to Cmax (Tmax) of Cobimetinib
Description: Plasma samples for determination of Cobimetinib concentration were collected prior to dosing and at 2, 4, 6 and 24 hours after dosing on Days 1 and 21 of Cycle 1. The sampling will allow determination of Tmax.
Time Frame: Pre-dose, 2, 4, 6, and 24 hours post-dose on Cycle 1 Days 1 and 21 (pre-dose=within 4 hours prior to dose; cycle length=28 days)
Population: as for outcome 18
Measure: Median (Full Range); unit: hr
Arm/Group | Phase I (Tablet) Cobimetinib (0.6 mg/kg) | Phase I (Tablet) Cobimetinib (0.8 mg/kg) | Phase I (Tablet) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (0.6 mg/kg) | Phase I (Suspension) Cobimetinib (0.8 mg/kg) | Phase I (Suspension) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (1.33 mg/kg) | Phase II (Suspension) Cobimetinib (1 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 5 | 12
hr
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 5 | 6 | 6 | 7 | 8 | 4 | 9
  Cycle 1 Day 1 | 4 [2 to 6] | 2 [2 to 6] | 3 [2 to 4] | 4 [2 to 6] | 4 [2 to 6] | 2 [2 to 4] | 5 [2 to 6] | 4 [2 to 6]
  Cycle 1 Day 21: number analyzed (Participants) | 5 | 5 | 5 | 6 | 6 | 8 | 2 | 9
  Cycle 1 Day 21 | 4 [2 to 6] | 4 [2 to 6] | 2 [2 to 4] | 4 [2 to 6] | 2 [2 to 4] | 3 [2 to 6] | 4 [4 to 4] | 2 [2 to 6]

20. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to 24 Hours (AUC0-24) of Cobimetinib
Description: Plasma samples for determination of Cobimetinib concentration were collected prior to dosing and at 2, 4, 6 and 24 hours after dosing on Days 1 and 21 of Cycle 1. The sampling will allow determination of AUC0-24.
Time Frame: as for outcome 19
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Phase I (Tablet) Cobimetinib (0.6 mg/kg) | Phase I (Tablet) Cobimetinib (0.8 mg/kg) | Phase I (Tablet) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (0.6 mg/kg) | Phase I (Suspension) Cobimetinib (0.8 mg/kg) | Phase I (Suspension) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (1.33 mg/kg) | Phase II (Suspension) Cobimetinib (1 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 5 | 12
hr*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 8 | 3 | 9
  Cycle 1 Day 1 | 865 (83.0) | 1006 (100) | 1432 (50.0) | 743 (67.4) | 1111 (144) | 1627 (74.0) | 1567 (33.1) | 589 (79.5)
  Cycle 1 Day 21: number analyzed (Participants) | 5 | 5 | 5 | 6 | 6 | 8 | 2 | 9
  Cycle 1 Day 21 | 836 (83.5) | 2802 (111) | 2382 (38.4) | 1624 (80.4) | 1805 (109) | 2562 (104) | 2511 (104) | 1402 (59)

21. Secondary Outcome: Apparent Clearance (CL/F) of Cobimetinib
Description: Plasma samples for determination of Cobimetinib concentration were collected prior to dosing and at 2, 4, 6 and 24 hours after dosing on Days 1 and 21 of Cycle 1, and within 4 hours prior to dosing on Day 1 of Cycle 2.
Time Frame: Pre-dose, 2, 4, 6, and 24 hours post-dose on Cycle 1 Days 1 and 21; pre-dose on Cycle 2 Day 1 (pre-dose=within 4 hours prior to dose; cycle length=28 days)
Population: Please note that for this Outcome Measure, the Apparent Clearance of Cobimetinib could not be calculated/estimated as PK samples were collected only up to 24hr post dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Phase I (Tablet) Cobimetinib (0.6 mg/kg) | Phase I (Tablet) Cobimetinib (0.8 mg/kg) | Phase I (Tablet) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (0.6 mg/kg) | Phase I (Suspension) Cobimetinib (0.8 mg/kg) | Phase I (Suspension) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (1.33 mg/kg) | Phase II (Suspension) Cobimetinib (1 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 5 | 12
L/hr | NA (NA) — The Apparent Clearance of Cobimetinib could not be calculated/estimated as PK samples were collected only up to 24hr post dosing which resulted in insufficient data to calculate CL/F. | NA (NA) — The Apparent Clearance of Cobimetinib could not be calculated/estimated as PK samples were collected only up to 24hr post dosing which resulted in insufficient data to calculate CL/F. | NA (NA) — The Apparent Clearance of Cobimetinib could not be calculated/estimated as PK samples were collected only up to 24hr post dosing which resulted in insufficient data to calculate CL/F. | NA (NA) — The Apparent Clearance of Cobimetinib could not be calculated/estimated as PK samples were collected only up to 24hr post dosing which resulted in insufficient data to calculate CL/F. | NA (NA) — The Apparent Clearance of Cobimetinib could not be calculated/estimated as PK samples were collected only up to 24hr post dosing which resulted in insufficient data to calculate CL/F. | NA (NA) — The Apparent Clearance of Cobimetinib could not be calculated/estimated as PK samples were collected only up to 24hr post dosing which resulted in insufficient data to calculate CL/F. | NA (NA) — The Apparent Clearance of Cobimetinib could not be calculated/estimated as PK samples were collected only up to 24hr post dosing which resulted in insufficient data to calculate CL/F. | NA (NA) — The Apparent Clearance of Cobimetinib could not be calculated/estimated as PK samples were collected only up to 24hr post dosing which resulted in insufficient data to calculate CL/F.

ADVERSE EVENTS:
Time Frame: Baseline up until 30 days after the last dose of study drug (up to 5 years, 2 months)
Arm/Group | Phase I (Tablet) Cobimetinib (0.6 mg/kg) | Phase I (Tablet) Cobimetinib (0.8 mg/kg) | Phase I (Tablet) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (0.6 mg/kg) | Phase I (Suspension) Cobimetinib (0.8 mg/kg) | Phase I (Suspension) Cobimetinib (1 mg/kg) | Phase I (Suspension) Cobimetinib (1.33 mg/kg) | Phase II (Suspension) Cobimetinib (1 mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/8 | 0/5 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 2/6 | 2/6 | 1/7 | 2/8 | 2/5 | 5/12
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6 | 7/7 | 8/8 | 5/5 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (Tablet) Cobimetinib (0.6 mg/kg) (N=6) | Phase I (Tablet) Cobimetinib (0.8 mg/kg) (N=6) | Phase I (Tablet) Cobimetinib (1 mg/kg) (N=6) | Phase I (Suspension) Cobimetinib (0.6 mg/kg) (N=6) | Phase I (Suspension) Cobimetinib (0.8 mg/kg) (N=7) | Phase I (Suspension) Cobimetinib (1 mg/kg) (N=8) | Phase I (Suspension) Cobimetinib (1.33 mg/kg) (N=5) | Phase II (Suspension) Cobimetinib (1 mg/kg) (N=12)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (Tablet) Cobimetinib (0.6 mg/kg) (N=6) | Phase I (Tablet) Cobimetinib (0.8 mg/kg) (N=6) | Phase I (Tablet) Cobimetinib (1 mg/kg) (N=6) | Phase I (Suspension) Cobimetinib (0.6 mg/kg) (N=6) | Phase I (Suspension) Cobimetinib (0.8 mg/kg) (N=7) | Phase I (Suspension) Cobimetinib (1 mg/kg) (N=8) | Phase I (Suspension) Cobimetinib (1.33 mg/kg) (N=5) | Phase II (Suspension) Cobimetinib (1 mg/kg) (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (7) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Iris hamartoma (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Precocious puberty (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid skin dryness (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic atrophy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic disc disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serous retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced transiently (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual field defect (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (7)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 1 (2)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (3) | 3 (5) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 4 (17) | 5 (8) | 4 (6) | 2 (3) | 4 (6) | 4 (10) | 4 (11)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 2 (7) | 3 (5) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4) | 4 (9) | 2 (2) | 2 (9) | 4 (7) | 2 (2) | 7 (14)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 3 (5) | 2 (2) | 2 (3) | 3 (3) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (2) | 1 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 3 (5)
Xerosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scarlet fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in ear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Anion gap increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood chloride increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 4 (8)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Body temperature decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cortisol decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (4)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mean cell volume increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (5)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (9) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (8)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (6) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 3 (4) | 2 (2) | 2 (4) | 3 (8) | 4 (4) | 3 (5) | 7 (11)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inappropriate affect (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal ulcer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sputum decreased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (6) | 1 (2) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 1 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pityriasis alba (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02639546/Prot_SAP_000.pdf